CLINICAL TRIAL: NCT01975870
Title: A stAPP to a Healthier Lifestyle: a Randomized Controlled Trial
Brief Title: A stAPP to a Healthier Lifestyle
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: Ministry of the Flemish Community (Other Government)
Responsible Party: Principal Investigator, Christophe Delecluse, Dr Professor Christophe Delecluse, Universitaire Ziekenhuizen KU Leuven
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: S55635
Record Dates: First submitted 2013-08-28; First posted 2013-11-05 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Sedentary Lifestyle
Keywords: Sedentary behavior, smartphone, application
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- intervention group (Experimental): use of application on smartphone for lifestyle counseling
  Interventions: Other: Application on smartphone
- control group (No Intervention): no use of application on smartphone

INTERVENTIONS:
Other: Application on smartphone — innovative application on smartphone which helps to increase the awareness of sedentary behavior of the user by messages, scoring system, ...
  Arms: intervention group

SUMMARY:
The main objective of the project is to make participants aware of their sedentary behavior (prolonged sitting behavior) and then to encourage behavioral change through the use of an innovative and fun application on a smartphone.

DETAILED DESCRIPTION:
Recent scientific research has shown that prolonged sitting, also called sedentary behavior may have adverse effects on health. An increased negative association was found with cardio-metabolic risk factors, type 2 diabetes and premature mortality.

The occurrence of these adverse health effects even appears to be independently of the degree of physical activity. There is more and more evidence to interrupt prolonged sitting regularly.

Until today there is still no international scientific standard that specifies how often the sitting behavior should be interrupted. Moreover, it is also unclear how long the breaks should take to counter adverse health effects. Only a few studies examined the health effects after an intervention that aimed to reduce the sitting behavior.

Currently, there is a great need for interventions in which one is made aware of the problem of sedentarity, but by which, one is equally encouraged changing behavior in the short as well as long term. In the proposed project the investigators therefore contribute to a good method to fight sedentary behavior in an innovative way. The investigators will try to achieve that goal through the development and implementation of an application on the smartphone.

Recent figures show that it is impossible to ignore the existence of the smartphone with all its applications. In 2011 40.4% of the Flemish people owned a smartphone. In the same year 650 000 smartphones were sold in Belgium. In 2012, according to projections this number should be increased by 250% to 1.625 000.

The smartphone is a very popular tool that can be used for the adoption of a healthy lifestyle. There are meanwhile a lot of sport and exercise apps that measure physical activity (eg Runkeeper Pro or Fitness Builder) and give more information around physical activity. Motion sensors, which are standard built-in in a smartphone, are often used for this purpose.

In the development of the app and the associated processes in this project, the principles of Self Determination Theory (SDT) are taken into account. This theoretical framework makes it possible to aim for a change in behavior in the short and in the long term.

During the development of the app, the investigators respect the sense of autonomy, competence and social connectedness of the user. Recent research showed already that applications which generate awareness and at regular intervals supply reminders, and this while autonomy and trust in their own competencies are respected, are effective in reducing sedentary behavior.

The effectiveness of the application will be investigated by means of a controlled intervention study. In this study, a control- and intervention group of 30 participants are included.

At the beginning of the project, both the intervention group and the control group will fill in some scientific questionnaires about sedentary behavior (pre-test).

1. st week: During one week, both the control- and the intervention group will wear an activity monitor (ActivPal). In this way, the investigators can determine the degree of physical activity and sedentary behavior.
2. nd week: After this week, the control group is asked not to change lifestyle. The persons of the control group still wear the activity monitor. The intervention group can use the app for a week and at the same time the persons of the intervention group have to carry the activity monitor. They can choose how they use the application (as they prefer, depending on the profile eg no advice versus daily advice received).

After the 2nd week, both the control and the intervention group are invited and fill in the questionnaire (post-test). Data from the activity monitor are retrieved. Now the investigators can examine if sedentary behavior of the intervention group was significantly decreased by the use of the app, compared to the sedentary behavior of the control group. Moreover, the investigators will also examine whether the way of use of the app (cfr profile) has an effect on the result.

ELIGIBILITY:
Inclusion Criteria:

* age between 19-59 years
* participants must own a smartphone
* participants have a sedentary lifestyle (prolonged sitting attitude)

Exclusion Criteria:

* people with mobility problems

Ages: 19 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2013-09; Primary Completion 2014-06 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Change in sedentary behavior | Pre measurements after first week, post measurements after second week
  Objective sedentary behavior: measured by ActivPal (monitor) Subjective sedentary behavior: measured by subjective questionnaire

SECONDARY OUTCOMES:
Usability application | Post measurement after second week
  Subjective questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Delecluse, Prof Dr, Study Director — KU Leuven
Locations (1):
- KU Leuven, Leuven, Flemish Brabant, Belgium

REFERENCES:
- [Result] Owen N, Healy GN, Matthews CE, Dunstan DW. Too much sitting: the population health science of sedentary behavior. Exerc Sport Sci Rev. 2010 Jul;38(3):105-13. doi: 10.1097/JES.0b013e3181e373a2. PMID 20577058
- [Result] Dunstan DW, Howard B, Healy GN, Owen N. Too much sitting--a health hazard. Diabetes Res Clin Pract. 2012 Sep;97(3):368-76. doi: 10.1016/j.diabres.2012.05.020. Epub 2012 Jun 9. PMID 22682948
- [Result] Healy GN, Dunstan DW, Salmon J, Cerin E, Shaw JE, Zimmet PZ, Owen N. Breaks in sedentary time: beneficial associations with metabolic risk. Diabetes Care. 2008 Apr;31(4):661-6. doi: 10.2337/dc07-2046. Epub 2008 Feb 5. PMID 18252901
- [Result] Rutten GM, Savelberg HH, Biddle SJ, Kremers SP. Interrupting long periods of sitting: good STUFF. Int J Behav Nutr Phys Act. 2013 Jan 2;10:1. doi: 10.1186/1479-5868-10-1. PMID 23281722
- [Result] Swartz AM, Squires L, Strath SJ. Energy expenditure of interruptions to sedentary behavior. Int J Behav Nutr Phys Act. 2011 Jun 27;8:69. doi: 10.1186/1479-5868-8-69. PMID 21708007
- [Result] Ryan RM, Deci EL. Self-determination theory and the facilitation of intrinsic motivation, social development, and well-being. Am Psychol. 2000 Jan;55(1):68-78. doi: 10.1037//0003-066x.55.1.68. PMID 11392867